CLINICAL TRIAL: NCT05448248
Title: A Registry Study of Cerebral Venous Sinus Thrombosis in China
Brief Title: Multicenter Registry Study Of Cerebral Venous Thrombosis In China (RETAIN-CH)
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Collaborators: Brain Hospital of Hunan Provincial (Unknown); The First Affiliated Hospital of Zhengzhou University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Guizhou Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Capital Medical University, Capital Medical University
Other Study IDs: RETAIN-CH
Record Dates: First submitted 2022-07-02; First posted 2022-07-07 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Vein Thrombosis; Cerebral Venous Sinus Thrombosis
Keywords: Cerebral Venous Sinus Thrombosis
MeSH Terms: conditions — Intracranial Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will investigate the epidemiology, risk factors, diagnostics, treatment, and the long-term prognosis of cerebral venous thrombosis in China.

DETAILED DESCRIPTION:
The epidemiology, risk factors, diagnosis and treatment of Cerebral Venous Thrombosis (CVT) in China are still unclear. A retrospective hospital-based study will be conducted at fifty different hospitals across 31 provinces in China. This study will use ICD-10 to search patients diagnosed with CVT between January 1, 2018 and June 15, 2022 across 31 provinces and municipalities of 104 hospitals in China. Risk factors, clinical and radiological findings, treatment and short-term outcomes will be recorded from the hospital record system. Finally, a prospective follow-up will be conducted for all of the patients enrolled above. By combining data collected from retrospective hospital records with the new follow-up, it will be possible to better understand the epidemiology, risk factors, diagnosis, treatment and the long-term prognosis of CVT in China.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral venous sinus thrombosis, deep cerebral vein thrombosis and cortical vein thrombosis diagnosed by digital subtraction angiography (DSA), magnetic resonance venography (MRV), computed tomography venography (CTV) or high-resolution magnetic resonance imaging (HR-MRI).

Exclusion Criteria:

* None of the patient, trustee or immediate family members signed the informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cerebral venous sinus thrombosis, deep cerebral vein thrombosis and cortical vein thrombosis.
Sampling Method: Probability Sample
Enrollment: 3276 (Actual)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Favorable clinical outcome (modified Rankin score 0-1) | Baseline to three years
All-cause mortality | Baseline to three years
  A combination of death form of all causes

SECONDARY OUTCOMES:
Recurrence of cerebral venous thrombosis | Baseline to three years
  Diagnosed by DSA, MRV, CTV or HR-MRI
Favorable clinical outcome (modified Rankin score 0-2) | Baseline to three years
Headache after CVT | Baseline to three years
  Headache Impact Test - 6 score
Incidence of hemorrhagic complication | Baseline to three years
  Extracranial hemorrhage (fall in hemoglobin of 2 gram/dl or more within 48 hours) or intracranial hemorrhage
Recanalization rate of cerebral venous system | Baseline to three years
Incidence of epilepsy | Baseline to three years
Incidence of acute ischemic stroke | Baseline to three years
Incidence of pulmonary embolism | Baseline to three years
Psychological distress after CVT | Baseline to three years
  Population Health Questionnaire (PHQ)-9 score

CONTACTS AND LOCATIONS:
Locations (1):
- Xuan Wu Hospital，Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Bian H, Wang X, Liu L, Yan F, Lu S, Hui W, Zhou C, Duan J, Li M, Chen J, Meng R, Cao L, Wang L, Ji X. Multicenter registry study of cerebral venous thrombosis in china (RETAIN-CH): Rationale and design. Brain Behav. 2024 Apr;14(4):e3353. doi: 10.1002/brb3.3353. PMID 38622893